CLINICAL TRIAL: NCT01544231
Title: Plasma Neutrophil Gelatinase Associated Lipocalin (NGAL) Levels During Emergency Management of Rhabdomyolysis: Predicting Renal Failure
Brief Title: Plasma Neutrophil Gelatinase Associated Lipocalin Levels During Emergency Management of Rhabdomyolysis
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-I/2011/SP-03; 2011-A01059-32 (Other: RCB number)
Record Dates: First submitted 2012-02-23; First posted 2012-03-05 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-12

CONDITIONS: Rhabdomyolysis; Acute Kidney Failure
Keywords: Neutrophil Gelatinase Associated Lipocalin; predicting acute kidney failure; emergency room
MeSH Terms: conditions — Rhabdomyolysis; Acute Kidney Injury; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Adult patients with suspected rhabdomyolysis admitted to the participating University Hospital emergency rooms (see inclusion/exclusion criteria).
  Interventions: Biological: Plasma NGAL level

INTERVENTIONS:
Biological: Plasma NGAL level — The plasmatic level of Neutrophil Gelatinase Associated Lipocalin is measured in ng/ml/

SUMMARY:
This research project consists of a prospective diagnostic study conducted on patients with clinical suspicion of rhabdomyolysis admitted to the emergency rooms of the University Hospitals of Nimes, Montpellier, Paris, Nice and Toulon Inter Army Hospital. The main objective of this study is to determine whether the plasma level of Neutrophil Gelatinase Associated Lipocalin (NGAL) may be retained as a predictor of acute renal failure (ARF) occurring within 48 hours after admission for rhabdomyolysis.

DETAILED DESCRIPTION:
The secondary objectives of this are:

* to study plasma NGAL levels on admission to the emergency ward as a marker of morbidity and mortality by considering the following factors: duration of hospitalization, need for extracorporeal blood purification, ICU admission, death.
* to study the delay between the onset of the proposed cause of rhabdomyolysis and treatment initiation
* to study the delay between treatment initiation and the occurrence of ARF.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient hospitalized with Creatine Phospho-Kinase > 1000 UI/l

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Chronic renal insufficiency with dialysis
* The patient has an acute coronary syndrome
* Nephrotoxic medications within 72 hours prior to admission
* Need for a procedure involving the injection of iodine
* Patient in shock
* Occurrence of acute renal failure can be explained by a cause other than rhabdomyolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected rhabdomyolysis admitted to the participating University Hospital emergency rooms (see inclusion/exclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12-09 (Actual); Study Completion 2015-12-09 (Actual)

PRIMARY OUTCOMES:
Plasma NGAL level | Admittance to the ermergency room (ie at baseline)
  ng/ml

SECONDARY OUTCOMES:
Delay between initiation of treatment and beginning of acute renal failure | Day 2
  meaured in hours
Delay between cause and treatment | Day 2
  Hours elapsed between proposed cause of rhabdomyolysis and treatment initiation measured in hours.
Need for extracorporeal blood purification | Hospital discharge (expected average of 2-3 days)
  yes/no
Patient admitted to ICU? | Hospital discharge (expected average of 2-3 days)
  yes/no
Length of hospitalization | Hospital discharge (expected average of 2-3 days)
  measured in days
Patient deceased during hospitalization | Hospital discharge (expected average of 2-3 days)
  yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Pommet, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (5):
- France (5):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nice - Hôpital St-Roch, Nice
  - APHP - Groupe Hospitalier Pitié-Salpetrière, Paris
  - Hôpital Interarmées Sainte Anne, Toulon

REFERENCES:
- [Result] Pommet S, Coisy F, Demattei C, Balaguer L, de Bauwere DP, Grau-Mercier L, Markarian T, Bobbia X, Genre Grandpierre R. Does serum neutrophil gelatinase-associated lipocalin level predict acute kidney injury in patients with acute rhabdomyolysis in the emergency department? A multicentre prospective study. BMJ Open. 2024 Nov 17;14(11):e088859. doi: 10.1136/bmjopen-2024-088859. PMID 39551581